CLINICAL TRIAL: NCT00763139
Title: Inflammation and Insulin Resistance in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Associate Director of the Division of Clinical Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: P60AR056116 (NIH); P60AR056116 (NIH)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo First (Experimental): Placebo for first 8 weeks, then washout period for 4 weeks, and finally pioglitazone for 8 weeks.
  Interventions: Drug: Pioglitazone; Drug: Placebo
- Pioglitazone First (Experimental): Pioglitazone for first 8 weeks, then washout period for 4 weeks, and finally placebo for 8 weeks.
  Interventions: Drug: Pioglitazone; Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 45 mg by mouth once a day for 8 weeks
  Other Names: Actos
Drug: Placebo — By mouth once a day for 8 weeks

SUMMARY:
Rheumatoid arthritis (RA) is a form of arthritis that causes pain, swelling, stiffness, and loss of function in the joints. Over time, joint deformity, joint destruction, and loss of function can occur. Current treatment aims to improve symptoms, but there is no cure for the disease. Pioglitazone is drug that is effective in treating people with diabetes. This study will determine whether pioglitazone can also be used to effectively treat people with RA.

DETAILED DESCRIPTION:
RA is an autoimmune disease that causes long-term inflammation of the joints and sometimes other body tissues, too. Recent studies have found that there is an increased prevalence of coronary artery atherosclerosis, metabolic syndrome, and insulin resistance among people with RA. Furthermore, insulin resistance, which can lead to hyperinsulinemia-too much insulin in the blood-has been associated with RA disease activity and the severity of coronary artery atherosclerosis. These correlations suggest that inflammation and hyperinsulinemia somehow interact and facilitate one another.

Pioglitazone is a prescription drug that reduces insulin resistance and is currently used to treat people with diabetes. This study will determine whether pioglitazone can also be used to effectively treat people with RA. Specifically, the study will evaluate the effect of pioglitazone on inflammation, insulin resistance, and atherosclerosis.

Participation in this study will last about 20 weeks. At an initial 1-hour screening, participants will undergo a physical examination, medical history review, blood sampling, and, if female, a urine pregnancy test. Eligible participants will then return for the first of six monthly study visits. At this first visit, participants will be randomly assigned to receive either pioglitazone or placebo, both of which will be taken daily for 8 weeks. This will be followed by a 4-week wash-out period, during which no study treatments will be taken. Then, at Week 12, participants will begin daily treatments of whatever they were not assigned to originally. This second treatment phase will also last for 8 weeks.

All of the study visits will involve the same tests and procedures. The morning before each study visit, participants will collect their urine in a jug, which they will bring to the clinic. Participants will then undergo blood sampling, blood pressure measurements, and artery stiffness measurements. During the study visits at Weeks 4, 8, 16, and 20, participants will be asked to report on their symptoms, pain, and any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets the American College of Rheumatology (ACR) criteria for the diagnosis of rheumatoid arthritis (RA)
* Stable disease activity, as evidenced by no change in immunomodulating or anti-inflammatory therapy in the 1 month before study entry
* Moderate disease activity, as reflected by a minimum of three swollen and tender joints
* If female of childbearing potential, willing to use effective method of contraception

Exclusion Criteria:

* Allergic to pioglitazone
* Active cancer (other than skin cancer)
* HIV infected
* Currently receiving dialysis
* Received an organ or bone marrow transplant
* Heart failure
* Severe edema, as judged by the principal investigator
* Diabetes mellitus requiring drug therapy: levels of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than twice the upper limit of normal
* Underwent major surgery in the 3 months before study entry
* Severe comorbid condition that is likely to compromise survival or study participation
* Currently receiving gemfibrozil or rifampin
* Osteoporosis and not receiving osteoporosis medications
* Unwillingness, or other inability, to cooperate with study procedures
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Stein, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Clinical Research Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Ormseth MJ, Oeser AM, Cunningham A, Bian A, Shintani A, Solus J, Tanner S, Stein CM. Peroxisome proliferator-activated receptor gamma agonist effect on rheumatoid arthritis: a randomized controlled trial. Arthritis Res Ther. 2013;15(5):R110. doi: 10.1186/ar4290. PMID 24020899
- [Derived] Ormseth MJ, Oeser AM, Cunningham A, Bian A, Shintani A, Solus J, Tanner SB, Stein CM. Reversing vascular dysfunction in rheumatoid arthritis: improved augmentation index but not endothelial function with peroxisome proliferator-activated receptor gamma agonist therapy. Arthritis Rheumatol. 2014 Sep;66(9):2331-8. doi: 10.1002/art.38686. PMID 24782291

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo 1st, Pioglitazone 2nd: Placebo for first 8 weeks, then washout period for 4 weeks, and finally pioglitazone for 8 weeks.
  Pioglitazone: 45 mg by mouth once a day for 8 weeks
  Placebo: By mouth once a day for 8 weeks
- Pioglitazone 1st, Placebo 2nd: Pioglitazone for first 8 weeks, then washout period for 4 weeks, and finally placebo for 8 weeks.
  Pioglitazone: 45 mg by mouth once a day for 8 weeks
  Placebo: By mouth once a day for 8 weeks
Period: Overall Study
Arm/Group | Placebo 1st, Pioglitazone 2nd | Pioglitazone 1st, Placebo 2nd
Started | 17 | 17
Completed | 12 | 14
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — med change not allowed by protocol | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics of Participants: participants who met American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA), age 18 or older, with moderate disease activity and no change in immunomodulating or anti-inflammatory therapy in past month
Arm/Group | Baseline Characteristics of Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score Based on 28-joint Disease Activity Score (DAS28)
Description: A measure of disease activity based upon tender joint count of 28 joints, swollen joint count of 28 joints, erythrocyte sedimentation rate, and global disease activity (GH) as reported by participant. Calculation is as follows: DAS28=0.56*sqrt(t28) + 0.28*sqrt(sw28) + 0.70*Ln(ESR) + 0.014*GH
Time Frame: Measured after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pioglitazone Phase Baseline: All participants who took pioglitazone in phase one or phase 2 of the study were combined to compare to the placebo phase. Baseline results are reported here.
- Pioglitazone Phase After 8 Weeks: All participants who took pioglitazone in phase one or phase 2 of the study were combined to compare to the placebo phase. Results after 8 weeks are reported here.
- Placebo Phase Baseline: All participants who took placebo in phase one or phase 2 of the study were combined to compare to the pioglitazone phase. Baseline results are reported here.
- Placebo Phase wk 8/20: All participants who took placebo in phase one or phase 2 of the study were combined to compare to the pioglitazone phase. Results after 8 weeks are reported here.
Arm/Group | Pioglitazone Phase Baseline | Pioglitazone Phase After 8 Weeks | Placebo Phase Baseline | Placebo Phase wk 8/20
Number analyzed (Participants) | 34 | 34 | 34 | 34
units on a scale | 4.40 (1) | 4.03 (1.15) | 4.57 (1.28) | 4.48 (1.20)

2. Primary Outcome: Homeostasis Model Assessment (HOMA) for Insulin Sensitivity
Description: Homa is a measure of insulin sensitivity, using glucose measured in mmol/L and insulin measured in milliUnits per liter (mU/L) Calculated using the formula Glucose * Insulin/22/5
Time Frame: Measured after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pioglitazone Phase After 8 Weeks: All participants who took pioglitazone in phase one or phase 2 of the study were combined to compare to the placebo phase. Results after 8 weeks on medication are reported here.
Arm/Group | Pioglitazone Phase Baseline | Pioglitazone Phase After 8 Weeks | Placebo Phase Baseline | Placebo Phase wk 8/20
Number analyzed (Participants) | 34 | 34 | 34 | 34
units on a scale | 2.83 (2.5) | 2.44 (2.08) | 2.38 (1.75) | 3.11 (3.47)

3. Secondary Outcome: C-reactive Protein (CRP)
Time Frame: Measured after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Placebo Phase wk After 8 Weeks: All participants who took placebo in phase one or phase 2 of the study were combined to compare to the pioglitazone phase. Results after 8 weeks on medication are reported here.
Arm/Group | Pioglitazone Phase Baseline | Pioglitazone Phase After 8 Weeks | Placebo Phase Baseline | Placebo Phase wk After 8 Weeks
Number analyzed (Participants) | 34 | 34 | 34 | 34
mg/dl | 8.1 (11.41) | 5.02 (7.64) | 7.7 (13.6) | 8.25 (10.32)

4. Secondary Outcome: ESR
Description: sed rate
Time Frame: baseline and after 8 weeks on either placebo or pioglitazone
Measure: Mean (Standard Deviation); unit: mm/hr
Groups:
- Placebo Phase After 8 Weeks: All participants who took placebo in phase one or phase 2 of the study were combined to compare to the pioglitazone phase. Results after 8 weeks are reported here.
Arm/Group | Pioglitazone Phase Baseline | Pioglitazone Phase After 8 Weeks | Placebo Phase Baseline | Placebo Phase After 8 Weeks
Number analyzed (Participants) | 34 | 34 | 34 | 34
mm/hr | 18.5 (18.2) | 17 (17.06) | 19.5 (20) | 18.88 (20.8)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over the course of the 20 week study.
Groups:
- Pioglitazone: participants who met ACR criteria for RA, age 18 or older, with moderate disease activity and no change in immunomodulating or anti-inflammatory therapy in past month, during the period they were taking pioglitazone
- Placebo: participants who met ACR criteria for RA, age 18 or older, with moderate disease activity and no change in immunomodulating or anti-inflammatory therapy in past month, during the period they were taking placebo
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 2/34
Other Adverse Events (participants affected / at risk) | 6/34 | 6/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=34) | Placebo (N=34)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — Placebo Arm: 2 participants became pregnant, one when placebo was first intervention given, one when placebo was 2nd intervention given
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=34) | Placebo (N=34)
liver function tests elevated (Hepatobiliary disorders) | 2 (2) | 1 (1)
ankle edema (General disorders) | 3 (3) | 2 (2)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Study relatively small, but efficiently designed. Crossover design has the advantage of comparing changes in the same patient and the disadvantage that subtle, undetected carryover effects may occur. 8 week drug exposure shorter than most trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No